CLINICAL TRIAL: NCT05649839
Title: Design of a Prototype Garment Adapted to Demented Elderly Subjects With Disturbing Behavioral Problems in the Management of Sphincter Disorders
Acronym: GERONESIE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2018_843_0053
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Adapted Garment Prototype; Elderly; Problem Behavior; Dementia; Sphincter Disorders
Keywords: adapted garment prototype; patient dignity; elderly; behavioral troubles; Dementia; sphincter disorders
MeSH Terms: conditions — Problem Behavior; Dementia | interventions — Clothing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional garment (Active Comparator)
  Interventions: Other: garment
- prototype garment (Experimental)
  Interventions: Other: garment

INTERVENTIONS:
Other: garment — patient randomized in the experimental arm will wear the specially designed garment

SUMMARY:
Alzheimer's disease and related disorders (ADRD) are diseases whose frequency is increasing in elderly subjects. Their evolution is marked by the occurrence, in addition to cognitive disorders, of increasingly disruptive behavioral disorders that interfere with their management, as well as impairment of basic functions, including the occurrence of sphincter disorders responsible for daytime and nighttime urinary and fecal incontinence. These disorders are present in more than 80% of LAM patients and are of multifactorial origin.

It is difficult to get patients to accept wearing the necessary protection. They tend to remove or tear them off. This can frequently lead to stressful situations of agitation and inappropriate behavior for patients and uncomfortable continence management for caregivers.

In order not to be forced to use heavy physical restraints or therapeutics that promote drowsiness so that the patient cannot remove his or her protections, the only effective response today is to wear a garment. Unfortunately, the ones that exist today are strictly functional and are worn at night.

The use of such garments, during the day, in this indication, is therefore a common and usual practice today.

This results in an ethical problem for the caregivers. Indeed, worn during the day, rompers give the impression to the latter that they show a devaluing, infantilizing or even degrading image of the elderly person. This practice, although common and accepted because it is the only recourse to physical and chemical restraints to preserve the cleanliness and presentation of elderly patients, could lead to an impaired dignity which could be badly experienced by their close circle of friends and family as well as by the carers and could also have an impact on the overall effectiveness of the care .

This is the first time that a multi-professional team integrating doctors, caregivers, occupational therapists and engineers have reflected on the design of a garment that meets the expectations of caregivers, patients and their families. The romper thus designed must be able to retain the aesthetic characteristics of a garment that meets the tastes of the elderly while respecting their dignity.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in a cognitive-behavioral unit or long-term care or residents of the EHPAD at the St-Victor center - CHU Amiens-Picardie,
* patients with behavioral and sphincter disorders justifying the prescription of a romper.
* signature of a consent exclusion criteria

Exclusion Criteria:

* No next of kin
* Patients in terminal palliative care
* Patients whose morphology does not allow the use of prototypes (no adapted size)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
variation of satisfaction score between both groups of patients | 6 months
  Satisfaction score will be measured with an home-made questionary. Higher scores for highest satisfactory. the questionary is composed of 10 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bloch F, Joron E, Boutalha S, Mekchoudi S, Claviere M. Design of a prototype of clothing for older persons with neurocognitive diseases with behavioural troubles interfering with the management of sphincter disorders. Disabil Rehabil Assist Technol. 2025 Apr;20(3):692-698. doi: 10.1080/17483107.2024.2404701. Epub 2024 Sep 18. PMID 40164140